CLINICAL TRIAL: NCT04634786
Title: The Association Between Central Serous Chorioretinopathy and the Obstructive Sleep Apnea
Brief Title: Association Between CRSA and OSA
Acronym: CRSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A02305-34
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Chorioretinopathy; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This goal of this study is to know the association between the central serous chorioretinopathy and the obstructive sleep apnea. Many studies have been done in order to assess the association between the central serous chorioretinopathy and obstructive sleep apnea and the results are always controverses actually.

ELIGIBILITY:
Inclusion Criteria:

* Central serous chorioretinopathy since 6 months at least
* Patients beyond 18 years old

Exclusion Criteria:

- All retina pathology will be excluded : diabetes with affected retina, maculopathy, retina central veinous oclusion, epithéliopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The central serous chorioretinopathy is defined by RSD (retinal serous detachment) located to the macula, it must be diagnosed since 6 months.
  Patients with central serous chorioretinopathy will undergo a Berlin Questions to assess the risks to have an obstructive sleep apnea.
  More over, we measure the choroid's thickness by using EDI OCT(Enhanced depth imaging optical coherence tomography) The survey and the measure of the choroid's thickness will be performed during an ophthalmology routing consultation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-08-06 (Estimated); Study Completion 2021-08-06 (Estimated)

PRIMARY OUTCOMES:
Association between central serous chorioretinopathy and the obstructive sleep apnea. | During 3 months we will collect the results of Berlin survey.
  Percentage of high risks of obstructive sleep apnea in patients affected by central serous chorioretinopathy in using the Berlin survey.
  The Berlin questions include 3 categories:
  The category 1 is positive if 2 answers are positive. The category 2 is positive if 2 answers are positive. The category 3 is positive if 1 answer is positive. Finally, if 2 categories are positive, the patient is considered as high risk of obstructive sleep apnea.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France